CLINICAL TRIAL: NCT02507128
Title: Effects of Glucagon Like Peptide-1 on No-reflow in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effects of Glucagon Like Peptide-1 on No-reflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Wei Ren, MD (Other)
Responsible Party: Sponsor-Investigator, Chen Wei Ren, MD, Dr., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 301xnk
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Liraglutide; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 group (Experimental): The treatment started 30 min before PCI with a dose of 1.8 mg liraglutide (the treatment was administered in the ambulance).
  Interventions: Drug: liraglutide
- Control group (Placebo Comparator): the treatment started 30 min before PCI with a dose of 1.8 mg placebo (the treatment was administered in the ambulance).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide were taken 30 min before PCI.
  Other Names: glucagon like peptide-1
  Arms: GLP-1 group
Drug: placebo — Placebo were taken 30 min before PCI.
  Arms: Control group

SUMMARY:
The investigators planned to evaluate the effects of liraglutide on no-reflow in patients with acute ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a major cause of mortality and morbidity. Primary percutaneous coronary intervention (PCI) is currently the most effective treatment strategy for AMI. Brisk thrombolysis in myocardial infarction (TIMI) grade 3 flow immediately after PCI in patients with AMI is associated with improved clinical outcomes compared with lower flow grades. However, myocardial reperfusion is suboptimal in many patients, mostly because of the 'no-reflow' phenomenon. No-reflow is defined as suboptimal myocardial reperfusion in part of the coronary circulation without angiographic evidence of mechanical vessel obstruction. To date, however, very few drugs have been shown to reverse established no-reflow.

Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose, and GLP-1 analogues were recently introduced for the treatment of acute myocardial infarction. GLP-1 has antioxidant and anti-inflammatory properties, and may protect endothelial function. Experimental studies have also revealed that GLP-1 or its analogues protect against reperfusion injury in pigs. Exenatide, a GLP-1 analogue, was reported to reduce reperfusion injury in patients with ST-segment elevation myocardial infarction. Similarly, liraglutide was reported to reduce cardiac rupture and infarct size and improve cardiac output in normal and diabetic mice. To date, however, there is no clinical evidence for the effects of liraglutide on no-reflow in patients with AMI. Therefore, the aim of this study was to evaluate the effects of liraglutide pretreatment on myocardial no-reflow of prime PCI in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

Patients with ST-segment elevation myocardial infarction were eligible for the study.

Exclusion Criteria:

Patients were excluded for the following reasons: unconscious at presentation; had cardiogenic shock, hypoglycaemia, or diabetic ketoacidosis; had a history of myocardial infarction, stent thrombosis, or renal insufficiency; or had previously undergone coronary artery bypass surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
a change in the prevalence of no-reflow | immediately after PCI
  The primary efficacy variable was the prevalence of no-reflow assessed immediately post procedure.

SECONDARY OUTCOMES:
a change in troponin T | immediately after PCI, at 1,3,5 days after PCI
  Secondary efficacy variable was troponin T level.
a change in high-sensitivity C-reactive protein (hsCRP) | immediately after PCI, at 1,3,5 days after PCI
  Secondary efficacy variable was high-sensitivity C-reactive protein level.
a change in superoxide dismutase (SOD) | immediately after PCI, at 1,3,5 days after PCI
  Secondary efficacy variable was superoxide dismutase level.

OTHER OUTCOMES:
differences in the incidences of treatment-emergent adverse events | immediately after PCI, at 1,3,5 days after PCI
  Treatment-emergent adverse events (TEAEs): hypoglycaemia, pancreatitis, thyroid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Gibson CM, Cannon CP, Murphy SA, Marble SJ, Barron HV, Braunwald E; TIMI Study Group. Relationship of the TIMI myocardial perfusion grades, flow grades, frame count, and percutaneous coronary intervention to long-term outcomes after thrombolytic administration in acute myocardial infarction. Circulation. 2002 Apr 23;105(16):1909-13. doi: 10.1161/01.cir.0000014683.52177.b5. PMID 11997276
- [Background] Rezkalla SH, Kloner RA. Coronary no-reflow phenomenon: from the experimental laboratory to the cardiac catheterization laboratory. Catheter Cardiovasc Interv. 2008 Dec 1;72(7):950-7. doi: 10.1002/ccd.21715. PMID 19021281
- [Background] Muller O, Trana C, Eeckhout E. Myocardial no-reflow treatment. Curr Vasc Pharmacol. 2013 Mar 1;11(2):278-85. PMID 23506504
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607